CLINICAL TRIAL: NCT06694493
Title: Factors Associated With Quality of Life in Chronic Low Back Pain: A Structural Equation Modelling Study
Brief Title: Factors Associated With Quality of Life in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Phd, Kutahya Health Sciences University
Other Study IDs: 2024-d
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low-back Pain (cLBP)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to identify and validate the factors that may affect quality of life in patients with chronic low back pain.

DETAILED DESCRIPTION:
Participants between the ages of 18-65, who are willing to participate in the study and have low back pain for more than 3 months will be included in the study. The necessary demographic information will be obtained with a data form. For the evaluation; Visual Analogue Scale (VAS), Tampa Kinesiophobia Scale, Fear-Avoidance Beliefs Questionnaire, Roland-Morris Disability Questionnaire, Beck Depression Scale, Self-Efficacy for Managing Chronic Disease 6-Item Scale, Coping Strategies Inventory Short Form (CSI-SF), Pain Catastrophising Scale, Pittsburgh Sleep Quality Index, Short Form - 36 (Quality of Life Questionnaire) will be used. The data obtained in the study will be entered into SPSS 17 package programme (Greasley, 2007). Minimum-maximum values, arithmetic mean and standard deviation will be used to evaluate numerical data, and frequency distributions and percentages will be used to summarise categorical data. The data of the study will be analysed using Analysis of Moment Structures (AMOS) statistical package programmes. In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having low back pain for more than 3 months
* Being between the ages of 18-65

Exclusion Criteria:

* History of surgery in the spinal region
* Rheumatoid arthritis
* Tumour
* Autoimmune disease
* Neurological disease
* Psychiatric or cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People between the ages of 18-65, who volunteered to participate in the study, and who had low back pain for more than 3 months will be included in the study.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute
  Visual Analogue Scale (VAS) will be used to assess the pain intensity of the patients. Patients will be given a paper with a 10 cm straight line with numbers between 0 and 10 on it and asked to score according to the severity of pain. 0 points will be given in the absence of pain and 10 points will be given in the most severe pain.
Tampa Kinesiophobia Scale | 5 minute
  The TKS is a 17-question scale and is used in acute and chronic low back pain, fibromyalgia and musculoskeletal injuries and whiplash-related disorders. The scale has a 4-point Likert scale (1= Strongly disagree, 4= Strongly agree). The total score is calculated after reversing items 4, 8, 12 and 16. The person receives a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia. The Turkish reliability study of the Tampa Kinesiophobia Scale was conducted by Yılmaz et al. (2011)
Fear-Avoidance Beliefs Questionnaire | 5 minute
  Fear Avoidance Beliefs Questionnaire consists of 16 questions. It has two subscales: physical activity and work. The physical activity section consists of 5 questions and the work section consists of 11 questions. The questionnaire is a 7-point Likert type scale. The answers to the questionnaire are between strongly disagree (0 points) and strongly agree (6 points). Items 1, 8, 13, 14 and 16 are not included in the scoring. The Physical Activity section can receive a minimum of 0 and a maximum of 24 points. The labour section can score a minimum of 0 and a maximum of 42 points. As the total score approaches 0, it is accepted that there is a decrease in fear-avoidance behaviour within the section, and as it approaches the maximum score, it is accepted that there is an increase in fear-avoidance behaviour. The Turkish reliability and validity study of the Fear-Avoidance Beliefs Questionnaire was conducted by Bingül et al.
Roland-Morris Disability Questionnaire | 5 minute
  Roland Morris Disability Questionnaire was published by Roland and Morris in 1983 (Roland & Fairbank, 2000). It consists of 24 questions about the person's perception of low back pain and related disability. It consists of physical ability/activity (15), sleep/rest (3), psychosocial (2), home management (2), eating (1) and pain frequency (1). Patients are asked to answer all questions 'yes/no'. Each 'yes' answer is scored as 1 and each 'no' answer is scored as 0. Total score for 24 questions is calculated. In this questionnaire, a high score indicates a bad score. The Turkish validation study of the Roland-Morris Disability Questionnaire was conducted by Küçükdeveci et al.
Beck Depression Scale | 5 minute
  The Beck Depression Scale is a self-report questionnaire that assesses the presence and severity of depressive symptoms. It consists of 21 items. Each item is scored on a four-point scale ranging from 0 (none) to 3 (severe). Total scores can vary between 0 and 63. The reliability and validity findings of the questionnaire adapted to Turkish have been obtained.
Self-Efficacy for Managing Chronic Disease 6-Item Scale | 3 minute
  Self-Efficacy for Managing Chronic Disease 6-Item Scale was developed by Lorig and colleagues in English in 2001 (Lorig, Sobel, Ritter, Laurent, & Hobbs, 2001). The scale is graded on a 10-point scale ranging from 'not at all confident' to 'completely confident'. The scale score is the average of 6 items. High scores indicate high self-efficacy. If more than 1 response is given to an item and the items are consecutive, the low score is included in the calculation. If 2 responses are not consecutive, this item is excluded from the calculation. In order to calculate the scale, at least 4 items must be answered. The Turkish version is a valid and reliable tool for assessing the perceived self-efficacy level of patients with chronic diseases.
Coping Strategies Inventory Short Form (CSI-SF) | 5 minute
  Coping Strategies Long Form is the short form developed by Carver (1997) after being revised. Coping Strategies Inventory Short Form consists of 28 questions and 14 subscales. Responses to each item are evaluated in the range of 1-4 points. The raw score that can be obtained from the subscales varies between 2-8.
Pain Catastrophising Scale | 5 minute
  The Catastrophising Pain Scale (PCS) is used to measure catastrophising in response to pain through 13 statements with four possible options from 1 'never' to 4 'always'. Higher scores indicate greater catastrophised pain. The Turkish validity study of the scale was conducted by Süren et al. (2014)
Pittsburgh Sleep Quality Index (PSQI) | 5 minute
  PSQI is a scale developed to evaluate sleep quality and sleep disturbance in a one-month period. PSQI consists of 24 questions in total. The first 18 questions answered by the participant himself/herself are used in the calculation of the PSQI total score and component scores. The 18 items included in the scoring are grouped into 7 components. Each item is evaluated in the range of 0-3 points. The sum of the seven component scores constitutes the result of the PSQI. The lowest score is zero and the highest score is 21. A high total score indicates poor sleep quality. The sleep quality of individuals with a total score of 5 and below is considered 'good', while the sleep quality of individuals with a score above 5 is considered 'poor'. The validity and reliability study of the PSQI was conducted by Agargun et al. (1996) in our country.
Short Form - 36 Quality of Life Questionnaire (SF-36) | 7 minute
  The Short Form - 36 Quality of Life Questionnaire (SF-36) is a general measure of health status, rather than measuring the outcomes of specific conditions. There is evidence that the SF-36 can be used to monitor musculoskeletal conditions. The SF-36 is a health-related quality of life questionnaire consisting of 8 scales (physical functioning, role limitations due to physical health problems, pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health). Responses to items are converted into scale scores from 0 (worst health) to 100 (best health). One physical and one mental summary health measure are derived from the 8 scales.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)